CLINICAL TRIAL: NCT04588740
Title: Inorganic Nitrate: Sex Differences in Muscle Contractile Function and Efficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jason Allen, Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 21983
Record Dates: First submitted 2020-10-01; First posted 2020-10-19 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: exercise; beet root juice; dietary nitrate; nitric oxide
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, cross-over design. This means that all subjects will complete both supplementation phases in a randomized order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dietary nitrate (Active Comparator): The active treatment, beetroot juice (BEET IT, James White Drinks, Ipswich, UK), contains 6.2mmol of inorganic nitrate. Participants will continue supplementation until they complete all testing visits.
  Interventions: Drug: concentrated beet root juice
- Placebo (Placebo Comparator): The placebo beet root juice is made by the same company (BEET IT, James White Drinks, Ipswich, UK) and contains no inorganic nitrate.
  Interventions: Drug: Placebo beet root juice

INTERVENTIONS:
Drug: concentrated beet root juice — On average, we will expect subjects to ingest the supplement for approximately 5 days minimum depending on their testing schedule. On each testing day subjects will be asked to consume the two bottles of either beetroot juice (BRJ) or Placebo 2.5 hours before testing time. Specifically, for female subjects, they will be asked to start their supplementation on day 1 of menses. On day 3-4 they will take the last 2 shots. Female subjects' wash-out period will go according to their menstrual cycle as we will be controlling for hormone fluctuation (low vs high estrogen phase) know to interact with nitric oxide physiology.
  Other Names: dietary inorganic nitrate
  Arms: Dietary nitrate
Drug: Placebo beet root juice — This will follow the same supplementation regime as explained above but this supplement taste and looks exactly the same as the nitrate-rich beet root juice. It is provided by the same company that produces the concentrated beet root juice shots (Beet It, UK)
  Other Names: placebo
  Arms: Placebo

SUMMARY:
Dietary inorganic nitrate, in the form of beet root juice, is a nutritional intervention, considered to be an exercise enhancer due to its capacity to increase Nitric Oxide (NO) bioavailability. Increasing NO bioavailability has been associated with improved mitochondrial respiration, muscle tissue perfusion and contractile function which may lead to improved exercise capacity. However, the majority of the literature is on male subjects. This limits the applicability of this supplement in females. Therefore, our project aims to determine sex-differences and the specific sex-response across the menstrual cycle of dietary nitrate supplementation on exercise efficiency, strength and fatigue resistance.

DETAILED DESCRIPTION:
Dietary inorganic nitrate is a nutritional intervention, considered to be an exercise enhancer due to its capacity to increase Nitric Oxide (NO) bioavailability. Increasing NO bioavailability has been associated with improved mitochondrial respiration, muscle tissue perfusion and contractile function which may lead to improved exercise capacity. The amount of research investigating the effects of beet root juice supplementation (which contains a high concentration of inorganic nitrate) on exercise responses has increased dramatically in the last 10 years-with over 150 studies in the literature. To date there are only 7 studies looking at exercise responses following inorganic nitrate supplementation specifically in females. Given the physiological differences between males and females studies looking into sex-differences and the specific sex-response are warranted.

The purpose of this study is to investigate whether dietary nitrate supplementation has different effects on muscle contractile function in males and females. We will assess muscle function during an isokinetic protocol where subjects will have to produce maximum efforts at three different torque development speeds (i.e. 180, 270 and 360). This will be followed with a fatigue protocol which will consist of intermittent voluntary contractions at 60% of their maximal voluntary contraction until exhaustion provided by research in the Sport Medicine - Kinesiology department. Thus, we will be able to distinguish the effect of dietary nitrate on contractile function and its capacity to delay fatigue in a sex-specific manner.

The hypothesis of this study is that there will be a group difference between males and females for change in peak power and time to exhaustion after consuming dietary nitrate (in the form of concentrated beetroot juice) for 5 days.

In order to test this hypothesis, we will recruit 24 healthy recreationally active individuals (12 females + 12 males) in a randomized, double-blind, placebo controlled, cross over design.

Specific Aim 1: Determine the sex-differences of the effect of dietary nitrate supplementation on peak power. We hypothesize that the males will have larger improvement in peak power following dietary nitrate.

Specific Aim 2: Determine the sex-differences of the effect of dietary nitrate on fatigue during an intermittent isometric fatigue protocol. We hypothesize that the females will have a greater improvement in fatigue resistance than males.

Specific Aim 3: Determine the sex-differences of the effect of dietary nitrate on oxygen consumption during sub maximal exercise.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants in good general health as assessed by the standard procedures described below and specifically meeting normal blood pressure range (systolic: 120-129, diastolic: 80-84) and normal BMI range (18.5-24.9)

  * Engaged in physical activity and/or recreational sport but not highly-trained, as assessed by the investigator in personal consultation and laboratory stress test.
  * No orthopedic limitations.

Exclusion Criteria:

* • Known pulmonary, cardiovascular or metabolic disease

  * Food allergies including phenylketonurea (PKU)
  * Regular use of dietary supplements within 6 months prior to the start of the study
  * Taking any dietary/sport supplements that could affect nitrate metabolism: Sport supplements containing the amino acids L-arginine, L-citrulline, beta-alanine, Creatine, Nitrate based pre-work out supplements
  * Blood donation within 3 months prior to the start of the study
  * Substance abuse within 2 years of the start of the study
  * Smokers
  * Hyper- or hypotension medication
  * Pregnant or lactating
  * Not having a regular menstrual cycle (minimum of 10-12 menses per year)
  * Stopped using a contraceptive method or started a new contraceptive method within 3 months.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Muscle function - Maximal knee extensor speed and power determined using isokinetic dynamometry | Male subjects (2 occasions)- It will be measured on day 5 of supplementation (placebo or nitrate). Female subjects (4 times) - It will be measured between days 3-5 and 10-15 of their menstrual cycle in two different cycles.
  This is an isokinetic (same speed over range of motion) strength test that will measure peak torque of the quadricep and hamstring (Nm/kg) and average power (W/kg). The testing protocol will be completed at three different speeds 180degrees/second, 270degrees/second and 360degrees/second.

SECONDARY OUTCOMES:
Oxygen consumption during a submaximal exercise | Male subjects (2 occasions)- It will be measured on day 5 of supplementation (placebo or nitrate). Female subjects (4 times) - It will be measured between days 3-5 and 10-15 of their menstrual cycle in two different cycles.
  Treatment differences (BR v PL) and sex differences (females vs males) in exercise economy (i.e. oxygen consumption) during a submaximal exercise bout (i.e. 75% Gas exchange threshold).
Time to exhaustion during a high intensity exercise bout on a cycle ergometer | Male subjects (2 occasions)- It will be measured on day 5 of supplementation (placebo or nitrate). Female subjects (4 times) - It will be measured between days 3-5 and 10-15 of their menstrual cycle in two different cycles.
  Treatment differences (BR v PL) and sex differences (females vs males) in exercise capacity during a constant work rate (i.e. 70% delta) tested on a cycle ergometer.

CONTACTS AND LOCATIONS:
Overall Officials: Jason D. Allen, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this RCT, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.